CLINICAL TRIAL: NCT04979676
Title: Changing the Course of Social Anxiety in Adolescence: What Works, Why, and for Whom
Brief Title: Changing the Course of Social Anxiety in Adolescence
Acronym: TeenSAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Paula Vagos, Principal investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTDC/PSI-ESP/29445/2017; POCI-01-0145-FEDER-029445 (Other Grant/Funding Number: Fundo Europeu de Desenvolvimento Regional)
Record Dates: First submitted 2021-07-15; First posted 2021-07-28 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Adolescence; Therapeutic Change; Therapeutic Efficacy; Therapeutic Processes
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This work uses a randomized and parallel clinical trial methodology (although the different parallel conditions are collected sequentially over the duration of the trial) to assess the effectiveness of three therapeutic approaches (i.e., CT, CFT and ACT) with adolescents with SAD, compared to a waiting-list control group.
  Originally, participants were to be sequentially and over time recruited and allocated to the different parallel conditions (i.e., assignment to CT or to a wait-list control condition in the first year; assignment to CFT or to a wait-list control condition in the second year, and assignment to ACT in the third year). However, the Covid-19 pandemic forced us to adapt the interventions to an online individual format thus delaying the assignment to the experimental conditions. So, all participants recruited in the first year were assigned to the wait-list control group and later randomly allocated to an experimental condition by the responsible investigator.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator is unaware of which participants are allocated to which condition; she is only aware of the inclusion criteria all participants must fulfill. The investigator and outcome assessor/data analyst are also unaware of treatment outcome and blind to the allocation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Therapy (Experimental): Experimental group subjected to active individual psychotherapy based on developing skills relating to flexibility of attention, which in turn sustains adolescents adopting a more realistic perspective on social events and acting based on external (and not only internal) social information. Assessed weekly during the intervention period on symptom change. Also assessed at pre-intervention, post-intervention (i.e., 10 to 12 weeks later), 12-weeks follow, and 24-weeks follow-up.
  Interventions: Behavioral: Cognitive Therapy
- Compassion-focused Therapy (Experimental): Experimental group subjected to active individual psychotherapy based on developing skills relating to flexibility of attention, which in turn sustains adolescents adopting a more realistic perspective on social events and acting based on external (and not only internal) social information. Assessed weekly during the intervention period on symptom change. Also assessed at pre-intervention, post-intervention (i.e., 10 to 12 weeks later), 12-weeks follow, and 24-weeks follow-up.
  Interventions: Behavioral: Compassion-focused Therapy
- Acceptance and Commitment Therapy (Experimental): Experimental group subjected to active individual psychotherapy based on developing skills for acceptance, defusing, and focusing on the present moments, which in turn sustain acting in social events in line with ones valued actions instead of prioritizing the avoidance of negative internal experiences). Assessed weekly during the intervention period on symptom change. Also assessed at pre-intervention, post-intervention (i.e., 10 to 12 weeks later), 12-weeks follow, and 24-weeks follow-up.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Waiting-list control (Placebo Comparator): Group of participants with a main dignosis os social anxiety disorder not subjected to any psychological intervention within the current trial. Assessed at time 0, then at time 1 ten to twelve weeks after time 1, then again at time 3 twelve weeks later, and then again at time 4 another twelve weeks later (i.e., 24 weeks after time 1).
  Interventions: Behavioral: Cognitive Therapy; Behavioral: Compassion-focused Therapy; Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Cognitive Therapy — Experimental psychotherapy based on the cognitive model for social anxiety disorder, applied individually and remotely to participants fulfilling inclusion criteria.
  Other Names: CT@TeenSAD
  Arms: Cognitive Therapy; Waiting-list control
Behavioral: Compassion-focused Therapy — Experimental psychotherapy based on the principles of the compassion-focused model, applied individually and remotely to participants fulfilling inclusion criteria.
  Other Names: CFT@TeenSAD
  Arms: Compassion-focused Therapy; Waiting-list control
Behavioral: Acceptance and Commitment Therapy — Experimental psychotherapy based on the principles of the acceptance and commitment model, applied individually and remotely to participants fulfilling inclusion criteria.
  Other Names: ACT@TeenSAD
  Arms: Acceptance and Commitment Therapy; Waiting-list control

SUMMARY:
Social anxiety often reaches its peak during adolescence and may hold a noteworthy impact both at the social and academic levels. Though some adolescents easily learn to adequately cope with it, others become overwhelmed by social fears and end up avoiding social events or facing them with intense suffering. Adolescents with social anxiety disorder (SAD) seldom seek professional help and often become adults with SAD, making it necessary to timely intervene during early stages of the disorder and determine what works better, why, and for whom when trying to change the course of social anxiety in adolescence. Cognitive therapy (CT) has been the treatment of choice for adult SAD, but research within adolescent samples is scarce. More recently, third-wave cognitive approaches, namely compassion-focused therapy (CFT) and acceptance and commitment therapy (ACT), have also proven effective in treating mental disorders, but their efficacy towards adolescents' SAD remains unclear.

This research project intended to evaluate and compare the therapeutic efficacy of CT, CFT, and ACT as applied to adolescents with SAD, in comparison with waiting-listed, after intervention and over a 12-weeks and a 24-weeks follow-up, using a randomized parallel trial approach. This methodology will allow to test if intervened subjects diverge from the non-intervened SAD subjects, and if therapeutic change differs across intervention conditions. Therapeutic change process will be investigated, specifically if efficacy is mediated by change in the core constructs of each theoretical framework. Finally, moderators of change such the initial level of symptomology will be examined, as to determine which intervention works best for whom. The same procedures will be repeated for each intervention condition, namely recruitment, intervention, and assessment.

This research will provide evidence on which form of therapy may be the optimal choice in to intervene in SAD in general, and when dealing with diverse specific vulnerabilities associated with social fears. It will also add to the field of empirically validated therapies, with a specific focus on adolescence. From a societal perspective, the project will assist in empowering schools to contribute to shape how their students act and develop into socially apt adults.

DETAILED DESCRIPTION:
Social anxiety is characterized by emotional reactivity to social events in which individuals believes they can be subject to the scrutiny of others. Although normative during adolescence, along with the growing importance attributed to acceptance and integration with peers, it can come to fulfill criteria for social anxiety disorder (SAD; McNeil, 2010), which is an intense and disabling experience for adolescents (Rao et al., 2007). SAD refers to excessive and persistent fear of being evaluated in social interactions, also with peers, which leads to those situations being faced with high levels of suffering or, if possible, avoided (APA, 2013). If not subject to specialized intervention, SAD usually has a chronic course and is associated with the emergence of other psychiatric disorders (Essau et al., 2004). In Portugal, it is estimated about 8% of adolescents in the community meet criteria for SAD, including intense anxiety and frequent avoidance of social situations, as well as severe impairment of academic and social functioning and quality of life. Most of these adolescents (roughly 94%) did not seek or were referred to specialized intervention (Vagos et al., 2021), which points to the importance of offering acceptable, practical, and effective forms of intervention for PAS.

With adults, the treatment of choice for SAD is Cognitive Therapy (CT; Mavranezouli et al., 2015) derived from the model by Clark and Wells (1995). This model proposes that social anxiety is maintained by cognitive biases (i.e., negative automatic thinking and self-focused attention) that support the practice of safety or avoidance behaviors, so that the intervention is aimed at making the focus of attention more flexible in order to be able to invest in and be exposed to social situations and extract evidence from them that may help adjust one's own thoughts and social expectations. Based on a review of evidence of the presence of various components of this model also in adolescents, Leigh and Clark (2018) propose that it could be applicable to the understanding and intervention in SAD in adolescents, contributing to better therapeutic results. In fact, previous work supports the therapeutic effectiveness (Leigh et al., 2021; Leigh & Clark, 2016) and applicability of this approach in different contexts (Creswell et al., 2021; Leigh et al., 2021).

While cognitive therapy focuses on modifying the cognitive content elicited by self-focused attention during social events as a means of preventing safety and/or avoidance behaviors in these situations (Clark & Wells, 1995), third-generation therapies (i.e., Compassion-focused Therapy - CFT and Acceptance and Commitment Therapy - ACT) emphasize the modification of the way the person relates to these cognitive contents. CFT proposes that this relationship be based on a compassionate attitude, given that psychopathology is based on a relationship with one's own internal experiences that is excessively critical and punishing, also in children and adolescents (Carona et al., 2017). There is previous evidence pointing to the association between self-compassion and social anxiety in adults (Werner et al., 2012) and adolescents (Gill et al., 2012), as well as to the effectiveness of CFT for SAD in adults (Boersma al., 2018; Gharraee et al., 2018). As for ACTC, its application with adolescents is also conceived, assuming that psychopathology results from an avoidant relationship with ones' own negative internal experiences (Hallibturton & Cooper, 2015). Still, along with the scant evidence linking its core constructs (i.e., psychological flexibility) to social anxiety, research on the efficacy of this intervention for SAD is scarce, although pointing to promising results with adults (Dalrymple, & Herbert, 2007; Khoramnia et al., 2020; Ossman et al., 2006). The applicability of these therapies to SAD in adolescence remains to be elucidated.

In view of the above, evidence on the efficacy of the therapeutic offer for SAD in adolescence is still scarce. So, it is relevant to explore the therapeutic results of CT, CFT and ACT, as well as to explore the mechanisms by which each one enables change and with whom it can be most effective. Previous research has pointed to the importance of changing core constructs in the CBT intervention with adults with SAD (e.g., Santoft et al., 2019), but evidence regarding the therapeutic approaches under study is scarce. In addition, and considering the relevance of the intervention being adjusted to the characteristics of the person receiving the intervention (Beck et al., 2010), it is important to explore the moderators of therapeutic change, namely with regard to the severity of symptoms within what is proposed to be the main psychological vulnerability for each of the approaches under analysis.

The present work used a parallel clinical trial methodology (although different parallel conditions were collected sequentially over time) to assess the efficacy of three therapeutic approaches (i.e., CT, CFT and ACT) with adolescents with SAD, compared to a waiting list control group, and using four data collection times (i.e., pre-intervention/time 0, post-intervention/time 1, 12-weeks follow-up/time3, and 24-month follow-up/time 4). All participants included in the waiting-list control group were offered the opportunity to receive psychological intervention, after the waiting period. All procedures involved in this study (i.e., sampling, data collection to assess the efficacy of the intervention, and implementation of the intervention) were implemented after a positive position from the Ethics Committee of the institution hosting the investigation, authorization from the General Directorate of Education on the data collection protocol to be implemented, partnership with national secondary schools, authorization of legal guardians of adolescents, and consent of the adolescents themselves. Furthermore, this investigation complied with all applicable ethical and deontological requirements.

The sampling process included two phases. The first phase was the screening of participants. Collaboration protocols were established with 26 secondary schools so that all 10th and 11th grade students of a school were invited to fill out a self-report questionnaire that assesses social anxiety, thus contributing to homogeneity with regard to the age group and social and academic experiences of the potential participants. Students with scores on this questionnaire above the normative average in Portugal were invited to participate in an individual assessment through a semi-structured diagnostic interview, to verify compliance with the inclusion and exclusion criteria described elsewhere in this form. Having fulfilled these criteria, adolescents were invited to join the study and fill out selected primary and secondary outcome measures to assess the efficacy of the interventions. They were firstly allocated to the waiting list-control group; later, participants from the waiting-list as well as newly recruited participants were sequentially allocated to one of the intervention groups over time The waiting-list control group was recruited in the first year of the research. Fifty-two participants initially accepted to participate in the study, but only 41 adolescents responded to at least one assessment moment, with the other 11 refusing to participant before any assessment moment. The 41 participants were contacted at the four evaluation moments as stated above. Of these, 21 participants completed all assessment moments. Participants initially allocated to the waiting-list control condition (including the ones that did not complete the 4 assessment moments) were contacted to be re-evaluated in the beginning of the second year of the research. The ones still fulfilling the inclusion criteria were offered the possibility of receiving an intervention (i.e., of being allocated to an experimental condition). Of the 52 participants that initially accepted to participate in the study, we were able to contact and evaluate 30 of them - 28 still met criteria for inclusion in an experimental group, 1 did not present SAD symptoms and 1 was receiving psychological intervention. Of the 28 participants fulfilling inclusion criteria, 3 refused the intervention and 25 were randomly allocated to the CFT or CT condition (20 to the CFT and 5 to the CT condition), along with another newly recruited 20 participants (18 to the CT and 2 to the CFT interventions). At this moment, 22 participants had been allocated to the CFT condition (1 of which dropped out) and 23 were allocated to the CT condition (6 of which dropped out). At the end of the second year of the research project, 21 participants had completed the CFT intervention and 17 had completed the CT intervention. In the third year of the project 28 adolescents (3 screened in the second year of the project and 25 screened in the second year of the project) were recruited and assigned to the ACT and CT conditions (4 to the CT intervention and 24 to the ACT intervention) so that all conditions had the minimum number of participants necessary for data analysis. Two participants dropped out of the ACT condition. In total, 92 participants enrolled in the study. All participants in all conditions were followed and continue to be followed over the four defined moments. Additionally, participants were/will be evaluated to verify the presence or absence of SAD at the 24-month follow-up/time 4 using the same semi-structured diagnostic interview used to assess initial inclusion/exclusion criteria.

Interventions followed a structured brief manual (i.e., 10 weekly sessions and 2 booster sessions 1 and 2 months after the core program was completed) and were implemented in individual online format via videoconference, according to the time availability of each adolescent; the facilitator had adequate training in psychology and in the therapeutic approach to be implemented.

Collected data will be used to investigate the therapeutic efficacy of each for the experimental intervention conditions across the four assessment moments, on its own, in comparison with each other, and comparing to a waiting-list control condition. Psychotherapeutic efficacy is usually tested against waiting-list control groups, based on the assumption that if the intervention and control groups started similarly at pre-intervention and present differently at post-intervention, the intervention is responsible for the observed change. This procedure is well established in the literature but has seldom been applied to adolescent SAD or to the different theoretical approaches tackled in this trial. Processes of change will also be analyzed as reflected in therapeutic change in constructs that were considered transversal to the intervention (e.g., social anxiety) being mediated by change in core constructs for each intervention. In addition, the moderating effect of initial levels of interference and intensity of symptomatology will be explored across experimental intervention conditions.

ELIGIBILITY:
Inclusion criteria for all experimental and the control group are:

* Aged between 15 and 18 years old at screening phase;
* Self-reported intensity of social anxiety higher than that reported by a normative comparable sample (Cunha et al., 2004);
* Main diagnosis of Social Anxiety Disorder as evaluated via the Mini-Kid (Rijo et al., 2016).

Exclusion criteria for all experimental and the control group are:

* Psychotic symptoms or suicidal risk as assessed via the Mini-Kid (Rijo et al., 2016);
* Being part of the special needs teaching system;
* Currently receiving psychological intervention/counselling.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Social anxiety and Avoidance Scale for Adolescents - Anxiety scale | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess intensity of discomfort felt when: 1) Interacting in new social events, 2) Interacting with the opposite sex, 3) Interacting assertively, 4) Performing in formal social situations, 5) Performing in new social situations, and 6) Eating and drinking in public. Previous psychometric information indicates factorial validity for the six-factor measurement model via exploratory and confirmatory factor analyses, very good internal consistency values for all measures, convergent validity in relation to other measures of anxious and depressive symptoms, and measurement invariance across gender and age (Cunha et al., 2008; Vagos et al., 2013).
Change in Social anxiety and Avoidance Scale for Adolescents - Avoidance scale | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess frequency of avoidance of: 1) Interacting in new social events, 2) Interacting with the opposite sex, 3) Interacting assertively, 4) Performing in formal social situations, 5) Performing in new social situations, and 6) Eating and drinking in public. Previous psychometric information indicates factorial validity for the six-factor measurement model via exploratory and confirmatory factor analyses, very good internal consistency values for all measures, convergent validity in relation to other measures of anxious and depressive symptoms, and measurement invariance across gender and age (Cunha et al., 2008; Vagos et al., 2013).
Change in Sheehan disability scale | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess functional impairment caused by social anxiety symptomatology at three inter-related domains: school/ academic performance, social life, and family life. Has previously proved to be sensitive in discriminating the presence/ absence of psychopathology (Pinto-Gouveia et al., 2000).
Change in Clinical Global Impression Scale for Social Anxiety | Severity will be assessed at Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 Week 7, Week, 8, Week 9, Week 10, Week 34. Change will be assessed at Week 2, Week 3, Week 4, Week 5, Week 6 Week 7, Week, 8, Week 9, Week 10.
  Clinician report of social anxiety symptoms. Has previously shown construct validity in relation to self-reported and clinician-administered measures of social anxiety, depression, impairment, and quality of life (Zaider et al., 2003). Includes measures of severity and change.
Social Anxiety Session Change Index | Week 2, Week 3, Week 4, Week 5, Week 6 Week 7, Week, 8, Week 9, Week 10.
  Self-report instrument used to assess how participants in the experimental groups perceive to have changed since the beginning of treatment in level of anxiety in social/ performance events, in avoidance of those events, in concern about embarrassing or humiliating themselves, and in social anxiety related daily interference. Has previously shown adequate internal consistency, validity in relation to concurrent perceived change in fear of negative evaluation, validity in relation to social anxiety, and severity of symptoms and improvement as reported by the clinician (Hayes et al., 2008).
Change in diagnostic assignment | Baseline e week 34
  Participants were/will be evaluated to verify the presence or absence of SAD at the 24-month follow-up/time 4 using the same semi-structured diagnostic interview used to assess initial inclusion/exclusion criteria.

SECONDARY OUTCOMES:
Change in Safety Behaviors in Social Situations Scale for Adolescents | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess practice of safety behaviors in social situations. Has previously shown factorial validity of the one-factor measurement model via exploratory factor analyses, good internal consistency and temporal stability, construct validity in relation to measures of social anxiety, criterion validity in relation to the presence/ absence of social anxiety disorder, and sensitivity to therapeutic change (Silva et al., 2010).
Change in Social Thoughts and Beliefs Scale | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess negative automatic thoughts common in socially anxious individuals, pertaining to discomfort in social interactions and to discomfort in public performance. Has previously shown factorial validity of a two-factor measurement model via exploratory factor analyses, very good internal consistency for all measures, and convergent validity in relation to a measure of social anxiety (Vagos et al., 2010).
Change in Self-focused Attention Scale | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess focus of attention in social situations, namely focus of attention in one's behavior and focus of attention in one's physiological arousal. Has previously shown factorial validity of a two-factor measurement model via exploratory factor analyses and good to excellent internal consistency for both factors (Fontinho e Salvador, 2012).
Change in Self-compassion Scale for Adolescents | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess external shame. Has previously shown factorial validity of the one-factor measurement model via confirmatory analyses, very good internal consistency, measurement invariance across gender, convergent validity in relation to measures of depressive, anxious and stress symptoms, self-criticism and self-reassurance, and experiential avoidance (Vagos et al., 2016).
Change in Other as Shamer Scale - Brief for Adolescents | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess external shame. Has previously shown factorial validity of the one-factor measurement model via confirmatory analyses, very good internal consistency, measurement invariance across gender, convergent validity in relation to measures of depressive, anxious and stress symptoms, self-criticism and self-reassurance, and experiential avoidance (Vagos et al., 2016).
Change in Forms of self-criticizing/attacking & self-reassuring scale - Adolescents | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess self-criticism and the ability to self-reassure, by measuring perceptions of an inadequate self, of a reassured self, and of a hated self. Has previously shown factorial validity for the three-factor measurement model via principal component analysis followed by varimax rotation, acceptable to excellent internal consistency for all factors, and convergent validity in relation to measures of anxiety and depression (Silva e Salvador, 2011).
Change in Avoidance and Fusion Questionnaire for Youth | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess psychological inflexibility. Has previously shown factorial validity of the one-factor measurement model via confirmatory factor analyses, very good internal consistency and temporal stability, and construct validity in relation with acceptance/ mindfulness, depressive and anxious symptoms, and social self-concept and comparison (Cunha & Santos, 2011).
Change in Social Anxiety - Acceptance and Action Questionnaire | Baseline, Week 10, Week 22, Week 34.
  Self-report instrument used to assess experiential acceptance associated with social anxiety symptomatology as reflected in willingness to experience social anxiety symptoms and moving towards valued life directions despite social anxiety symptoms. Has previously shown factorial validity of the two-factor measurement model via confirmatory factor analyses, very good internal consistency and temporal stability, construct validity in relation to measures of social anxiety, of mindfulness/ acceptance, and other anxious and depressive symptoms, criterion validity in relation to the presence/ absence of social anxiety disorder (Martins et al., 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Psicologia e Ciências da Educação - Universidade de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as participants were guaranteed anonymity and confidentiality of their individual data. Datasets with alphanumerical identities given to each participant may be made available, either by publishing data or upon reasonable request directed at with the principal investigator.

REFERENCES:
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Washington, DC: Author.
- [Background] Beck C, McSweeney JC, Richards KC, Roberson PK, Tsai PF, Souder E. Challenges in tailored intervention research. Nurs Outlook. 2010 Mar-Apr;58(2):104-10. doi: 10.1016/j.outlook.2009.10.004. PMID 20362779
- [Background] Boersma, K., Håkanson, A., Salomonsson, E., & Johansson, I. (2014). Compassion Focused Therapy to counteract shame, self-criticism and isolation. A replicated single case experimental study for individuals with social anxiety. Journal of Contemporary Psychotherapy, 45(2), 89-98. https://doi.org/10.1007/s10879-014-9286-8
- [Background] Carona, C., Rijo, D., Salvador, M.C., Castilho, P., & Gilbert, P. (2018). Compassion-focused therapy with children and adolescents. BJPsych Advances, 23(4), 240-252. https://doi.org/10.1192/apt.bp.115.015420
- [Background] Clark, D. M., & Wells, A. (1995). A cognitive model of social phobia. In G. Heimberg, M. R. M. R. Liebowitz, D. Hope, & F. Scheier (Eds.), Social phobia: Diagnosis, assessment, and treatment (pp. 69-93). New York: The Guilford Press.
- [Background] Creswell C, Leigh E, Larkin M, Stephens G, Violato M, Brooks E, Pearcey S, Taylor L, Stallard P, Waite P, Reynolds S, Taylor G, Warnock-Parkes E, Clark DM. Cognitive therapy compared with CBT for social anxiety disorder in adolescents: a feasibility study. Health Technol Assess. 2021 Mar;25(20):1-94. doi: 10.3310/hta25200. PMID 33759742
- [Background] Cunha, M., Pinto-Gouveia, J.P., Alegre, S., & Salvador, M.C. (2004). Avaliação da ansiedade na adolescência: A versão portuguesa da SAS-A. Psychologica, 35, 249-263.
- [Background] Cunha, M., Pinto-Gouveia, J. P., & Salvador, M. C. (2008). Social fears in adolescence - The social anxiety and avoidance scale for adolescents. European Psychologist, 13(3), 197-213. https://doi.org/10.1027/1016-9040.13.3.1974
- [Background] Cunha, M. & Santos, A.M. (2011). Avaliação da inflexibilidade psicológica em adolescentes: Estudo das qualidades psicométricas da versão portuguesa do Avoidance and Fusion Questionnaire for Youth (AFQ-Y). Laboratório de Psicologia, 9, 133-146.
- [Background] Cunha, M., Xavier, A., & Vitória, I. (2013). Avaliação da auto-compaixão em adolescentes: Adaptação e qualidades psicométricas da Escala de Auto-Compaixão. Journal of Child and Adolescent Psychology, 4(2), 95-117.
- [Background] Dalrymple KL, Herbert JD. Acceptance and commitment therapy for generalized social anxiety disorder: a pilot study. Behav Modif. 2007 Sep;31(5):543-68. doi: 10.1177/0145445507302037. PMID 17699117
- [Background] Essau CA, Lewinsohn PM, Olaya B, Seeley JR. Anxiety disorders in adolescents and psychosocial outcomes at age 30. J Affect Disord. 2014 Jul;163:125-32. doi: 10.1016/j.jad.2013.12.033. Epub 2014 Jan 2. PMID 24456837
- [Background] Fontinho, A. & Salvador, M. C. (2012). O papel da atenção auto focada na fobia social na adolescência: validação da versão portuguesa da Escala de Atenção Auto Focada (SFA) e estudos preliminares [Unpublished master dissertation]. Faculty of Psychology and Educational Sciences of University of Coimbra.
- [Background] Gharraee, R., Rajrishi, K., Farani, A., Bolhari, J., & Farahani, H. (2018). A randomized controlled trial of compassion focused therapy for social anxiety disorder. Iranian Journal of Psychiatry and Behavioral Sciences, 12(4), e80945. https://doi.org/10.5812/ijpbs.80945
- [Background] Gill C, Watson L, Williams C, Chan SWY. Social anxiety and self-compassion in adolescents. J Adolesc. 2018 Dec;69:163-174. doi: 10.1016/j.adolescence.2018.10.004. Epub 2018 Oct 13. PMID 30326397
- [Background] Halliburton, A. & Cooper, L. (2015). Applications and adaptations of Acceptance and Commitment Therapy (ACT) for adolescents. Journal of Contextual Behavioral Science, 1-11. https://doi.org/10.1016/j.jcbs.2015.01.002
- [Background] Hayes SA, Miller NA, Hope DA, Heimberg RG, Juster HR. Assessing Client Progress Session by Session in the Treatment of Social Anxiety Disorder: The Social Anxiety Session Change Index. Cogn Behav Pract. 2008 May 1;15(2):203-2011. doi: 10.1016/j.cbpra.2007.02.010. PMID 25075171
- [Background] Khoramnia S, Bavafa A, Jaberghaderi N, Parvizifard A, Foroughi A, Ahmadi M, Amiri S. The effectiveness of acceptance and commitment therapy for social anxiety disorder: a randomized clinical trial. Trends Psychiatry Psychother. 2020 Jan-Mar;42(1):30-38. doi: 10.1590/2237-6089-2019-0003. PMID 32321083
- [Background] Leigh E, Clark DM. Cognitive Therapy for Social Anxiety Disorder in Adolescents: A Development Case Series. Behav Cogn Psychother. 2016 Jan;44(1):1-17. doi: 10.1017/S1352465815000715. Epub 2015 Dec 7. PMID 26640031
- [Background] Leigh E, Clark DM. Understanding Social Anxiety Disorder in Adolescents and Improving Treatment Outcomes: Applying the Cognitive Model of Clark and Wells (1995). Clin Child Fam Psychol Rev. 2018 Sep;21(3):388-414. doi: 10.1007/s10567-018-0258-5. PMID 29654442
- [Background] Leigh E, Creswell C, Stallard P, Waite P, Violato M, Pearcey S, Brooks E, Taylor L, Warnock-Parkes E, Clark DM. Delivering cognitive therapy for adolescent social anxiety disorder in NHS CAMHS: a clinical and cost analysis. Behav Cogn Psychother. 2021 Mar 1:1-13. doi: 10.1017/S1352465821000035. Online ahead of print. PMID 33645498
- [Background] Martins, M.J., Vieira, S., Salvador, M.C., Mackenzie, M.B., & Kocovski, M.L. (2015). Social anxiety - Acceptance and Action Questionnaire: Adaptation and validation in a Portuguese adolescent sample. Unpublished manuscript.
- [Background] Mavranezouli I, Mayo-Wilson E, Dias S, Kew K, Clark DM, Ades AE, Pilling S. The Cost Effectiveness of Psychological and Pharmacological Interventions for Social Anxiety Disorder: A Model-Based Economic Analysis. PLoS One. 2015 Oct 27;10(10):e0140704. doi: 10.1371/journal.pone.0140704. eCollection 2015. PMID 26506554
- [Background] McNeil, D.W. (2010). In. Hofmann, G. & DiBartolo, P.M. (Eds), Social anxiety: Clinical, developmental and social perspectives (pp. 3-21). Oxford, UK: Elsevier.
- [Background] Ossman, W. A., Wilson, K. G., Storaasli, R. D., & McNeill, J. R. (2006). A preliminary investigation of the use of acceptance and commitment therapy in group treatment for social phobia. International Journal of Psychology and Psychological Therapy, 6(3), 397-416.
- [Background] Pinto-Gouveia, J., Cunham M. & Salvador, M. (2000). Um protocolo para a avaliação clínica da fobia social através de questionários de auto-resposta. In J. Pinto-Gouveia (Ed.), Ansiedade Social: Da timidez à fobia social (pp. 237-258). Coimbra: Quarteto Editora.
- [Background] Rao PA, Beidel DC, Turner SM, Ammerman RT, Crosby LE, Sallee FR. Social anxiety disorder in childhood and adolescence: descriptive psychopathology. Behav Res Ther. 2007 Jun;45(6):1181-91. doi: 10.1016/j.brat.2006.07.015. Epub 2006 Sep 27. PMID 17007813
- [Background] Rijo D, Brazao N, Barroso R, da Silva DR, Vagos P, Vieira A, Lavado A, Macedo AM. Mental health problems in male young offenders in custodial versus community based-programs: implications for juvenile justice interventions. Child Adolesc Psychiatry Ment Health. 2016 Nov 1;10:40. doi: 10.1186/s13034-016-0131-6. eCollection 2016. PMID 27822300
- [Background] Silva, C., Salvador, M. C. (2011). A Escala das Formas de Auto-Criticismo e de Auto-Tranquilização (FSCRS): Características Psicométricas na População Adolescente [Poster Presentation]. II Jornadas Internacionais do CINEICC: Novos olhares sobre a mente, Coimbra, Portugal.
- [Background] Silva, S., Salvador, M. C., & Pinto-Gouveia, J. P. (2010). Escala de Comportamentos de Segurança em Situações Sociais para Adolescentes (ECSSSA): Características psicométricas. Poster presentation at I Jornadas de Iniciação à Investigação em Psicologia. Coimbra: CINEICC.
- [Background] Santoft F, Salomonsson S, Hesser H, Lindsater E, Ljotsson B, Lekander M, Kecklund G, Ost LG, Hedman-Lagerlof E. Processes in cognitive behavior therapy for social anxiety disorder: Predicting subsequent symptom change. J Anxiety Disord. 2019 Oct;67:102118. doi: 10.1016/j.janxdis.2019.102118. Epub 2019 Jul 27. PMID 31487573
- [Background] Vagos, P., Pereira, A., & Beidel, D.C. (2010). Adaptação e validação de uma escala de medida de cognição na ansiedade social. Avaliação Psicológica, 9(3), 393-402. https://doi.org/10.1037/a0019782
- [Background] Vagos, P., & Pereira, A., & Cunha, M. (2013). Evaluating social fears in late adolescence: Study with a Portuguese Sample. European Journal of Developmental Psychology, 11(3), 373-385. https://doi.org/10.1080/17405629.2013.841093
- [Background] Vagos, P., Ribeiro da Silva, D., Brazão, N., Rijo, D. & Gilbert, P. (2016). Dimensionality and measurement invariance of the Other as Shamer Scale across diverse adolescent samples. Personality and Individual Differences, 98, 289-296. https://doi.org/10.10167j.psid.2010.04.046
- [Background] Werner KH, Jazaieri H, Goldin PR, Ziv M, Heimberg RG, Gross JJ. Self-compassion and social anxiety disorder. Anxiety Stress Coping. 2012;25(5):543-58. doi: 10.1080/10615806.2011.608842. Epub 2011 Sep 6. PMID 21895450
- [Background] Zaider TI, Heimberg RG, Fresco DM, Schneier FR, Liebowitz MR. Evaluation of the clinical global impression scale among individuals with social anxiety disorder. Psychol Med. 2003 May;33(4):611-22. doi: 10.1017/s0033291703007414. PMID 12785463
- [Background] Vagos, P., Figueiredo, D., Miguel, R., Ganho, A., Rijo, D., Lima, L., & Salvador, M.C. (2021). Ansiedade social na adolescência em contexto escolar: Uma experiência (não tão) normativa [Social anxiety in adolescence in schools: A (not so) normative experience]. Poster presented at the XVI Congresso Internacional Galego-Português de Psicopedagogia.